CLINICAL TRIAL: NCT04364087
Title: Impact of Glucose Metabolism Abnormalities on Live Birth Rate in South-East Asian Women With Polycystic Ovary Syndrome
Brief Title: Glucose Metabolism and Live Birth Outcomes in PCOS
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 08/20/ĐĐ-BVMD
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: PCOS; Infertility; Diabetes; PreDiabetes
MeSH Terms: conditions — Infertility; Diabetes Mellitus; Prediabetic State | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile PCOS women: All Vietnamese, infertile women, diagnosed with PCOS according to the Rotterdam criteria (2003) at IVFMD Tan Binh and IVFMD Phu Nhuan will be enrolled to the study.
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Oral glucose tolerance test with 75 g glucose (75 g OGTT) will be performed to those with normal fasting glucose and HbA1C levels. Women will be recommended to have normal diet for 3 days and overnight fasting for at least 8 hours. The blood withdrawal will be performed twice: (i) fasting and (2i) 2 hours after solution administration. The volume of blood for each test is 2 ml. Impaired glucose tolerance will be diagnosed when two-hour glucose levels of 140 to 199 mg/dL (7.8 to 11.0 mmol/l) (American Diabetes Association, 2018).

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine and reproductive disorder in which insulin resistance (IR) is proposed as a key pathophysiological feature of the disease's symptoms and consequences. Diabetes and rediabetes, a significant consequence of IR, are related to a higher risk of diabetes mellitus, future cardiovascular events, and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
All Vietnamese infertile women with PCOS, according to the Rotterdam criteria present at IVFMD, will be enrolled in the study. Phenotypes of PCOS are classified into A, B, C, and D due to hyperandrogenism (HA), ovulatory dysfunction (OD), and polycystic ovarian morphology (PCOM)

* A: HA + OD + PCOM
* B: HA + OD
* C: HA + PCOM
* D: OD + PCOM

All patients enrolled in this study will have:

* Standard anthropometric data will be done by professional and experienced physicians according to standard study protocol: Weight, height, waist and hip circumference, waist-to-hip ratio, and BMI calculated, followed by World Health Organization guidelines for Asian women. Trained midwives evaluated hirsutism and acanthosis nigricans, and fat mass was measured in the abdomen area using specific calipers (Accu-Measure®).
* Gynecologic ultrasound scan
* Blood tests:

A fasting blood sample was obtained. Luteinizing hormone (LH) (with a coefficient of variation [CV] 2.3%), follicle-stimulating hormone (FSH) (CV 3.5%), estradiol (CV 2.7%), progesterone (CV: 6.2%), prolactin (CV: 5.2%), sex hormone binding globulin (SHBG) (CV 5.6%), total testosterone (CV 8.4%) were measured by Elesys technique, Cobas e411 system. FAI was calculated using the formula: FAI = serum testosterone in nmol/L/serum SHBG in nmol/L × 100. Thyroid stimulating hormone (TSH) (CV 6.0%), free thyroxin (fT4) (CV 5.05%) were measured by Access 2 immunoassay system. High-density lipoprotein cholesterol (HDL-C) (CV 2.4%), low-density lipoprotein cholesterol (LDL-C) (CV 2.0%), and triglyceride (CV 1.76%) were measured by Beckman Coulter AU480 system. Fasting serum insulin (CV 2.8%) was measured by Elesys technique, Cobas e411 system. The Homeostasis Model Assessment of Insulin Resistance Index (HOMA-IR) was used to estimate insulin sensitivity. HOMA-IR was calculated as FPG in mmol/L × fasting insulin in mIU/mL/22.5 (Matthews et al., 1985). A 2 mL blood sample was withdrawn and stored in a vacutainer with nature oxalate and EDTA additive.

- Glucose tests:

+ After a fast of ≥4 hours, FPG (CV 0.9%) was measured by Beckman Coulter AU480 analyzer, and HbA1c (CV 1.00%) were measured by Tosoh HLC-723GX analyzer; participants who had not fasted for ≥4 hours were asked to return for measurement of FPG the next day.

Diagnosis of diabetes mellitus will be made when fasting glucose ≥126 mg/dL (7 nmol/L) or HbA1C ≥6.5% (48 mmol/mol) (American Diabetes Association, 2018). When glucose ≥126 mg/dL (7 nmol/L) or HbA1C ≥6.5% (48 mmol/mol) (American Diabetes Association, 2018).

* Oral glucose tolerance test with 75 g glucose (75 g OGTT) will be performed on those with normal fasting glucose and HbA1C levels. Women will be recommended to have a normal diet for three days and overnight fasting for at least 8 hours. The blood withdrawal will be performed twice: (i) fasting and (2i) 2 hours after solution administration. The volume of blood for each test is 2 ml. Impaired glucose tolerance will be diagnosed when two-hour glucose levels of 140 to 199 mg/dL (7.8 to 11.0 mmol/l) (American Diabetes Association, 2018).

  - Hyperandrogenism:
* Clinical hyperandrogenism: Hirsutism using the modified Ferriman Gallwey score (mFG) and severe acne
* Biochemical hyperandrogenism: free testosterone (normal range below 2,53nmol/ml), free testosterone index, SHBG

Following the assessment of glucose metabolism, all patients identified with preconception glucose metabolism disorders (e.g., prediabetes or diabetes) were referred to endocrinologists for specialized preconception care. This included lifestyle modifications and/or pharmacological interventions, aiming to optimize metabolic health before conception and potentially reduce adverse pregnancy outcome. Conception was achieved through various methods, including natural conception, ovulation induction combined with intrauterine insemination (OI/IUI), or in-vitro fertilization/ in-vitro maturation (IVF/IVM). These treatment options were counseled based on the recommendations from the 2023 international evidence-based guideline, in which first-line therapy involves optimizing preconception health and lifestyle, followed by OI with letrozole. Timed intercourse was recommended in the absence of male factor infertility, while IUI was offered in cases with mild male factor. IVF/IVM was indicated after failure of these initial approaches. Final decisions were individualized through shared decision-making, depending on clinical indications and patient preference (Teede et al., 2023b). Pregnancy outcomes, including pregnancy rates, live births and pregnancy outcomes, were tracked and documented over a 24-month follow-up period from the time of study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Vietnamese women aged 18-40 years
* Diagnosed with polycystic ovary syndrome (PCOS) according to the Rotterdam criteria (2003)
* Having indications for infertility treatment

Exclusion Criteria:

* Thyroid-stimulating hormone (TSH) > 5 mIU/mL
* Serum prolactin (PRL) > 30 ng/mL
* History of hypothyroidism
* Cushing's syndrome
* Premature ovarian insufficiency
* Late-onset or non-classic congenital adrenal hyperplasia
* Any other concomitant endocrinopathy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile Vietnamese women aged 18-40 years, diagnosed with polycystic ovary syndrome (PCOS) according to the Rotterdam 2003 criteria, who present for infertility treatment at IVFMD.
Sampling Method: Non-Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate at 24 months following enrollment into the study | From enrollment until delivery (up to 24 months after enrollment)
  Live birth was defined as the delivery of a live infant after 22 weeks of gestation, regardless of the method of conception.

SECONDARY OUTCOMES:
Gestational diabetes mellitus | From enrollment until delivery (up to 24 months after enrollment).
  Diagnosis based on standard criteria recorded in medical records.
Hypertensive disorders of pregnancy | From enrollment until delivery (up to 24 months after enrollment).
  Includes gestational hypertension, preeclampsia, and eclampsia.
Miscarriage | From enrollment until delivery (up to 24 months after enrollment).
  Pregnancy loss before 22 weeks of gestation.
Preterm birth | From enrollment until delivery (up to 24 months after enrollment).
  Delivery before 37 completed weeks of gestation.
Birthweight | At delivery (up to 24 months after enrollment).
  Neonatal birthweight measured in grams at delivery; categorized as low birthweight (<2500 g) or macrosomia (≥4000 g).
Gestational age at birth | At delivery (up to 24 months after enrollment).
  Gestational age in completed weeks at delivery.
Neonatal Intensive Care Unit (NICU) admission | At delivery (up to 24 months after enrollment).
  Admission to NICU after birth (yes/no).
Neonatal respiratory distress | At delivery (up to 24 months after enrollment).
  Clinical diagnosis of respiratory distress requiring intervention.
Baseline glycemic status (diabetes, prediabetes, or normal glucose tolerance before infertility treatment) | At baseline (at enrollment, before treatment).
  Glycemic status will be determined before initiation of infertility treatment, based on the 75-g oral glucose tolerance test (OGTT), fasting plasma glucose, and HbA1c, according to the American Diabetes Association (ADA) 2023 criteria. Participants will be categorized into: Diabetes mellitus, Prediabetes, Normal glucose tolerance.
  Unit of Measure: Number of participants (%) in each category.

CONTACTS AND LOCATIONS:
Overall Officials: Lan TN Vuong, MS, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No